CLINICAL TRIAL: NCT07262840
Title: Facilitating Health Behavior Change in High-Risk Individuals for Colorectal Cancer: A Randomized Controlled Trial
Brief Title: Health Behavior Change in High-Risk Colorectal Cancer Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenna Qian, Doctoral Researcher, School of Nursing, China Medical University, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HBC-HR-CRC
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Health Behavior; Colorectal Neoplasms; Primary Prevention/Methods
Keywords: Health Promotion；Health Behavior；Lifestyle Intervention；High-Risk Population
MeSH Terms: conditions — Health Behavior; Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Promotion Lifestyle Intervention Group (Experimental): Participants in this arm receive a 12-week, multi-component health promotion program based on the Health Promotion Model. The intervention includes: 1) Five in-person group workshops focusing on knowledge, motivation, planning, and maintenance; 2) Online support via a WeChat group for daily behavioral check-ins (e.g., exercise, diet) and peer support; 3) Educational articles and resources; 4) Techniques from Motivational Interviewing and Acceptance and Commitment Therapy to foster psychological adjustment and behavior change.
  Interventions: Behavioral: Multi-component Health Promotion Lifestyle Intervention
- Standard Care (Active Comparator): Participants in this arm receive standard care, which may include general health information about colorectal cancer prevention. They do not participate in the structured workshops, online check-ins, or specialized support of the experimental intervention. They will complete all the same assessment questionnaires as the intervention group. They may be offered the intervention program after the study is complete (wait-list design).
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Multi-component Health Promotion Lifestyle Intervention — 1. Intervention Name:
     Multi-Component Health Promotion Lifestyle Intervention
  2. Description:
  This is a structured, theory-based intervention designed to facilitate health behavior change in individuals at high risk for colorectal cancer. It is distinguished by its foundation in the Health Promotion Model and the Integrative Model of Health Behavior Change, and its use of a blended online and offline delivery model over a 12-week period.
  The intervention is organized into five sequential modules:
  Cognitive Reconstruction: Provides essential knowledge about colorectal cancer (etiology, risk factors) and disease prevention strategies.
  Psychological Adjustment: Employs techniques from Motivational Interviewing to build intrinsic motivation and Acceptance and Commitment Therapy (ACT) to help participants manage distress and psychological barriers related to their cancer risk.
  Health Behavior Establishment: Guides participants in creating personalized health plans and builds self-effic
  Arms: Health Promotion Lifestyle Intervention Group
Other: Standard Care — Participants randomised to the control arm will receive standard care, which may include general health advice or publicly available educational pamphlets on colorectal cancer prevention. They will not receive any component of the structured multi-component health promotion lifestyle intervention (i.e., no group workshops, no WeChat-based check-ins, no psychological techniques training, and no facilitated peer support). However, they will be asked to complete all the same assessment questionnaires at the same time points as the intervention group. Upon completion of the final follow-up assessment, participants in this arm will be offered the opportunity to receive the full intervention program (wait-list design).
  Arms: Standard Care

SUMMARY:
Background Colorectal cancer is a significant health concern. For individuals identified as being at high risk for developing this disease, adopting healthy lifestyle behaviors is a powerful way to lower that risk. However, starting and maintaining these new habits can be challenging. This study aims to test a comprehensive support program designed to help high-risk individuals make and sustain these positive health behavior changes.

Purpose The main goal of this research is to see if a specially designed 12-week health promotion program can effectively help high-risk individuals improve their lifestyle (e.g., diet, exercise, smoking/alcohol use), increase their knowledge about colorectal cancer, and strengthen their confidence and motivation to stay healthy.

Study Groups Participants in this study will be randomly assigned (like flipping a coin) to one of two groups:

1. The Intervention Group: This group will take part in the 12-week health promotion program.
2. The Control Group: This group will receive general health information or standard care but will not participate in the special program.

Procedures The program for the Intervention Group includes:

* Educational Workshops: Five in-person group sessions to learn about cancer prevention, create personal health plans, and solve problems with others.
* Online Support: Regular health articles and tips sent through a private WeChat group.
* Daily Check-ins: Using the WeChat group for simple daily check-ins on exercise, fruit/vegetable intake, and smoking/alcohol use to build habit.
* Peer Support: Being paired with a "health buddy" and interacting with other participants for motivation.

All participants will be asked to complete several questionnaires at the beginning of the study, during the program, and after it ends (at 3 months) to measure their knowledge, beliefs, and lifestyle habits.

Duration The active program lasts for 12 weeks.

Potential Benefits Participants in the Intervention Group may benefit from improved health habits, a better understanding of how to reduce their cancer risk, and increased social support. Participants in the control group will receive general health information. If they wish, they will receive the same health materials and behavioral change intervention as the intervention group after the intervention concludes.

ELIGIBILITY:
Inclusion Criteria:

* Meets the criteria for being at high-risk for colorectal cancer as defined by the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Colorectal Cancer Screening and the relevant Chinese expert consensus on colorectal cancer diagnosis and treatment.
* Age ≥ 18 years.
* Has normal verbal communication and comprehension abilities.
* Provides informed consent and voluntarily agrees to participate in the study.

Exclusion Criteria:

* Has a prior diagnosis of any malignancy (cancer).
* Has a diagnosed severe psychiatric or psychological disorder.

Ages: 18 Months to 80 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Score change in the Health Promotion Lifestyle Scale for High-Risk Colorectal Cancer Population (HPLP-HRCP) | Baseline (Week 0), Post-intervention (Week 12)
  This is the primary outcome measure, assessed using the revised Health Promotion Lifestyle Profile for High-Risk Colorectal Cancer Population (HPLP-HRCP). This scale measures the level of health-promoting lifestyle behaviors. A higher total score indicates a better health-promoting lifestyle.

SECONDARY OUTCOMES:
Score change in Colorectal Cancer Knowledge Questionnaire (CRC-KQ) | Baseline (Week 0), Post-intervention (Week 12).
  Assessed using the 21-item Colorectal Cancer Knowledge Questionnaire. It consists of two dimensions: basic knowledge (15 items) and screening knowledge (6 items). Each correct answer scores 1 point. A higher total score indicates a higher level of colorectal cancer knowledge.
Score change in the Champion Health Belief Model Scale (CHBMS) | Baseline (Week 0), Post-intervention (Week 12).
  Assessed using the Chinese version of the Champion Health Belief Model Scale. It contains 36 items across 6 dimensions: perceived susceptibility, perceived severity, perceived benefits, perceived barriers, health motivation, and self-efficacy. A higher score on a 5-point Likert scale indicates stronger health beliefs toward adopting recommended health behaviors.
Score change in the Multidimensional Health Locus of Control Scale (MHLC) | Baseline (Week 0), Post-intervention (Week 12).
  Assessed using the Chinese version of the Multidimensional Health Locus of Control Scale. It has 18 items across 3 subscales (6 items each): Internal, Powerful Others, and Chance. Each subscale is scored from 6 to 36 on a 6-point Likert scale. A higher score on a subscale indicates a stronger tendency towards that specific locus of control.
Score change in the Kessler Psychological Distress Scale (K10) | Baseline (Week 0), Post-intervention (Week 12).
  Assessed using the Chinese version of the 10-item Kessler Psychological Distress Scale. Total scores range from 10 to 50. Higher scores indicate higher levels of psychological distress. Scores are categorized as: 10-15 (Well), 16-21 (Mild), 22-29 (Moderate), and 30-50 (Severe) distress.
Score change in the Perceived Social Support Scale (PSSS) | Baseline (Week 0), Post-intervention (Week 12).
  Assessed using the Chinese version of the Perceived Social Support Scale. It contains 12 items across 3 dimensions: family, friends, and significant others. Each item is rated on a 7-point Likert scale. A higher total score indicates a higher level of perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
What IPD will be shared? Individual participant data that underlie the results reported in the primary and secondary publications after de-identification. This will include demographic data, baseline characteristics, and all outcome measure scores (e.g., HPLP-HRCP, CRC-KQ, CHBMS, MHLC, K10, PSSS).
  When will IPD be available? Beginning 9 months after the publication of the main trial results and ending 36 months thereafter.
  Who can access the IPD?? Researchers who provide a methodologically sound proposal for use in an independent ethical review-approved meta-analysis or replication study.
  How can IPD be accessed? Proposals should be directed to the corresponding author via email. To gain access, requestors will need to sign a data access agreement. Data will be shared via a secure file transfer platform.
  What other documents will be available? The study protocol, statistical analysis plan, and informed consent form will be made available on ClinicalTrials.gov alongside the results.